CLINICAL TRIAL: NCT05155774
Title: Treatment Adherence With Twin-Blocks for Correction of Class II Malocclusion - a Randomized Controlled Trial on Two Check-up Prescriptions
Brief Title: Treatment Adherence With Twin-Blocks for Correction of Class II Malocclusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Jönköping County (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EPM 2017/382-31
Record Dates: First submitted 2021-11-02; First posted 2021-12-14 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-11

CONDITIONS: Compliance, Patient; Treatment Adherence
Keywords: Orthodontic; Removable; Compliance; Adherence; Twin Block
MeSH Terms: conditions — Patient Compliance; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessor will check outcome on blinded study models.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group, controlled every 6th week (Active Comparator): This group was controlled every 6th week, in accordance with what is deemed to be "golden standard" for treatment with a Twin Block orthodontic appliance.
  Interventions: Device: Twin block
- Test group, controlled every 4th week (Experimental): This group was controlled every 4th week, testing if a more frequent control interval would increase compliance with a Twin block orthodontic appliance.
  Interventions: Device: Twin block

INTERVENTIONS:
Device: Twin block — Twin Block orthodontic appliance for treating patients with Angle class II molar relationship and a large horizontal overjet, often in combination with an incomplete lip closure

SUMMARY:
To compare the effect of two control intervals (once every 4th week or once every 6th week) on the wear time of a Twin Block removable appliance.

DETAILED DESCRIPTION:
If the patient fulfill the inclusion criteria, they will be asked to participate in the study. After being informed about the study and the planned treatment, participants and their guardians will give their written consent to participate in the study.

Therafter they will be consecutively randomized into one of two groups with different control intervals, Group 1 (every 4th week) and Group 2 (every 6th week). They will recieve a clinical and radiological examination and then start treatment with a Twin Block appliance.

The Twin Block appliance will be fitted with a digital timer module to measure the wear time of the appliance objectively.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients (ASA 1 and 2)
* Overjet of 6 mm or more
* Incomplete lip closure

Exclusion Criteria:

* Severe chronic conditions such as asthma or allergies
* Neuroopsychiatric disorders
* Craniofacial syndromes
* Previous orthodontic treatment

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2020-10-22 (Actual)

PRIMARY OUTCOMES:
Wear time of the Twin Block appliance, compared between participants randomized into two groups with different check up intervals | From randomization to 12 months of treatment
  To measure if the wear time of the Twin Block appliance would increase if the control interval increased from once every 6th week to once every 4th week. The wear time was registered using the TheraMon system, and was measured in hours per day.

SECONDARY OUTCOMES:
Change in overjet, compared between participants randomized into two groups with different check up intervals | From randomization to treatment completion, up to 24 months.
  To see if change in overjet would differ between or within the groups before and after treatment was finished. Horizontal overjet was measured in millimetres on study casts before and after treatment was finished.
Change in overbite, compared between participants randomized into two groups with different check up intervals | From randomization to treatment completion, up to 24 months.
  To see if change in overbite would differ between or within the groups before and after treatment. Overbite was measured in millimetres on study casts taken before and after treatment.
Change in molar relationship, compared between participants randomized into two groups with different check up intervals | From randomization to treatment completion, up to 24 months.
  To see how molar relationship would be differ between or within the two groups before and after treatment, measured in Angle classification on study casts before and after treatment completion.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Magnusson, DDS, DMSc, Study Chair — Institute of Postgraduate Dental Education, department of Orthodontics, Jönköping, Sweden; Mikael Sonesson, DDS, DMSc, Study Chair — Orthodontic department, Faculty of odontology, Malmö University, Sweden
Locations (1):
- Institute of Postgraduate Dentaln Education, department of orthodontics, Jönköping, Jönköping City Council, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Depends on data security in europe and if the data can be securely shared in accordance with GDPR

REFERENCES:
- [Derived] Frilund E, Sonesson M, Magnusson A. Patient compliance with Twin Block appliance during treatment of Class II malocclusion: a randomized controlled trial on two check-up prescriptions. Eur J Orthod. 2023 Mar 31;45(2):142-149. doi: 10.1093/ejo/cjac046. PMID 35968672